CLINICAL TRIAL: NCT05577637
Title: Comparitive Study Between Uvb Phototherapy Alone and Uvb Photothearpy With Topical 0.03% Tacrolimus for Treatment of Vitiligo
Brief Title: Comparitive Study Between Uvb Alone and Uvb With Topical Tacrolimus 0.03% for the Treatment of Vitiligo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Rohida Rahmat, principle investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHAtd-26-Derm-22
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Vitiligo
Keywords: Phototherapy; tacrolimus; vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A topical tacrolimus 0.03% with uvb phototherapy (Active Comparator): Group A :contain 30 patients who have been treated with topical 0.03% tacrolimus twice daily at night and then received uvb phototherapy thrice weekly for 12 weeks
  Interventions: Drug: 0.03% tacrolimus twice daily was applied on group A patients with uvb phototherapy thrice daily
- Group B topical placebo twice daily with uvb phototherapy thrice weekly (Active Comparator): Group B :contain 30 patients received uvb phototherapy only thrice weekly for 12 weeks
  Interventions: Drug: 0.03% tacrolimus twice daily was applied on group A patients with uvb phototherapy thrice daily

INTERVENTIONS:
Drug: 0.03% tacrolimus twice daily was applied on group A patients with uvb phototherapy thrice daily — 0.03% tacrolimus twice daily was applied on group A patients with uvb phototherapy thrice daily
  Other Names: ointment eczemus

SUMMARY:
Vitiligo is a skin disorder that causes substantial social and psychological distress due to multiple patches of depigmentation.Disease can target at any age, but it appears to affect various parts of body due to loss of melanin. Although the exact cause of the disease is unknown, several theories suggest that genetic predisposition, autoimmunity, and increased vulnerability of melanocytes to the deleterious effects of harmful metabolites all play a role in disease causation. It impacts 0.1%-2% of the general population, with a 30% familial prevalence rate.

Vitiligo treatment still presents a therapeutic challenge for dermatologists despite a variety of therapeutic modalities. Topical steroids, ultraviolet B phototherapy (UVB 280nm-320nm), and photochemotherapy (PUVA i.e., psoralen plus UVA 329nm-400nm) are traditional treatment options. Topical calcipotriol and excimer laser are also used. According to research, narrowband UVB (NB-UVB) is effective when used alone.

Few studies, however also, have reported more than 75% re-pigmentation in patients treated with NB-UVB in conjunction with other modalities. Topical immunomodulators (tacrolimus, pimecrolimus) are considered safe and effective long-term treatments for vitiligo because they do not cause skin atrophy, which is associated with long-term use of topical corticosteroids. Tacrolimus is an effective treatment for vitiligo when used alone; in one study, 61% of patients showed more than 75% repigmentation when treated with tacrolimus alone. Another study found that when tacrolimus was combined with NB-UVB, 73% of patients experienced more than 50% repigmentation.

The objective of this research was to present a comparatively new mode of treatment that may be beneficial to vitiligo patients.

ELIGIBILITY:
Inclusion Criteria:

* patients having 20-60 years of age
* non pregnant
* no history of photosensitivity
* no history of immunosuppression or immunosuppressive drugs
* no histry of steroids use oral or topical in last four weeks

Exclusion Criteria:

* pregnancy
* lactation
* history of photosensitivity
* photo-aggravated dermatoses
* history of any immunosuppressive disorder or use of immunosuppressive medicine
* history of using steroids either oral or injectable within the previous one month
* history of skin malignancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
effectiveness of 0.03% topical tacrolimus with uvb phototherapy and placebo with uvb photothreapy is calculated through repigmentation using a formula {% re-pigmentation = Present % depigmentation ÷ Baseline % depigmentation x 100} | 12 weeks
  repigmentation assesed by {% re-pigmentation = Present % depigmentation ÷ Baseline % depigmentation x 100}

CONTACTS AND LOCATIONS:
Locations (1):
- cmh Abbottabad, Abbottabad, Khyber Pakhtunkhwa, Pakistan